CLINICAL TRIAL: NCT00204438
Title: Follicular Profiles After Administration of Oral Contraceptives at Different Times of the Follicular Phase of the Menstrual Cycle
Brief Title: Administration of Oral Contraceptives at Different Times of the Follicular Phase of the Menstrual Cycle
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Saskatchewan (Other)
Collaborators: Canadian Institutes of Health Research (CIHR) (Other Government)
Responsible Party: Principal Investigator, Roger Pierson, Ph.D. FEAS, FCAHS, MS, University of Saskatchewan
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: BMC 2001-249; CIHR MOP - 11489
Record Dates: First submitted 2005-09-12; First posted 2005-09-20 (Estimated); Last update posted 2016-11-28 (Estimated); Status verified 2016-11

CONDITIONS: Contraception
Keywords: female contraception; oral contraceptive; emergency contraceptive; ovary; follicle; ovulation
MeSH Terms: interventions — Desogestrel

INTERVENTIONS:
Drug: 0.15mg desogestrel /0.03mg ethinyl estradiol

SUMMARY:
We hypothesize that administration of OCs at varying follicular diameters will provide an appropriate model for the study of follicular atresia in women. Clinically, we hypothesize that the administration on OCs at different stages of the follicular phase will result in markedly different patterns of follicular development and/or atresia.

DETAILED DESCRIPTION:
This study is a single-centre, randomized, open-label, double-controlled protocol to study the patterns of ovarian follicular growth and regression in women administered 0.15mg desogestrel /0.03mg ethinyl estradiol at different stages of the follicular phase of the menstrual cycle.

We tracked the growth and regression of dominant follicles after administration of OC by means of highly sophisticated transvaginal ultrasonography and computerized image analysis techniques. The extremely high resolution ultrasonography of the ovarian follicles and the computer-assisted image analysis are unique to the Women's Health Imaging Research Laboratory (WHIRL) at the University of Saskatchewan. The synergyne (© R.A. Pierson) image analysis program was developed in the WHIRL and has the ability to allow assessment of the physiologic status of follicles as small as 6 to 10 mm. This unique protocol will allow us to characterize patterns of follicular growth and atresia under the suppressive effects of oral contraception, as well as the assessment of anovulatory follicles which may develop when OCs are administered at advanced stages of follicular development.

The working hypothesis is that the administration of monophasic OCs prior to and during the time of physiologic selection of the dominant follicle will prevent the development of an ovulatory follicle (selection occurs when the dominant follicle reaches 10mm [Baerwald & Pierson, unpublished data]). In addition, we hypothesize that administration of OCs after selection of the dominant follicle, at more advanced stages of follicular development will result in 1 of 4 scenarios: 1.) Ovulation of the dominant follicle, 2.) Regression of the dominant follicle, 3). Formation of a Hemorrhagic Anovulatory follicle (HAF) or Luteinized Unruptured Follicle (LUF), or 4.) Formation of a follicular cyst. We hypothesize that atresia of dominant follicles and formation of anovulatory follicular structures will be associated with limited endometrial development. In testing these hypotheses, we will determine if OCs can safely and effectively be administered at any time during the follicular phase of the menstrual cycle.

This study will evaluate the ovarian and uterine responses to administration of a combined dose of 0.15mg desogestrel /0.03mg ethinyl estradiol at 1 of 3 different stages of the follicular phase of the menstrual cycle. The objectives of the trial are to:

* Develop new and more user-friendly administration schemes for OC use;
* Use the administration of OCs at different stages of follicular development in women as a model for studying follicular atresia;
* Assess the differences in kinetics, physiologic status (state of viability or atresia), and ultrasonographic image attributes of follicles which grow, regress, ovulate, or form anovulatory follicular structures after the administration of exogenous steroid hormones;
* Assess endometrial response to ovarian suppression by ultrasonographic evaluation of endometrial thickness and endometrial pattern.

After screening measurements confirm subject eligibility, subjects will be randomized to initiate OC therapy at one of three different times of the menstrual cycle:

Experimental Group #1: receives OCs when the dominant follicle reaches 10mm Experimental Group #2: receives OCs when the dominant follicle reaches 14mm Experimental Group #3: receives OCs when the dominant follicle reaches 18mm

Fifteen women will be randomized to each of the 3 experimental groups in a stratified design scheme. Data collected from an ongoing OC trial (BMC# 2000-169) will serve as OC control data (n=15). Data collected from a previous study (BMC# 1988-80) will serve as natural cycle control data (n=60).

ELIGIBILITY:
Inclusion Criteria:

* Female volunteers of childbearing potential;
* Are first time users of OCs or have discontinued OCs at least 1 month prior to study entry;
* Aged between 18 and 35 years (extremes included);
* Normal body mass index (18-38);
* Has signed informed consent form;
* Is in good health as confirmed by medical history, physical examination, and PAP smear or colposcopy within the past 12 months with normal results.

Exclusion Criteria:

* Any contraindication for oral contraceptive use;
* Irregular menstrual cycles
* Ultrasonographic evidence of ovarian dysfunction, such as Polycystic Ovary Syndrome (PCOS);
* Pregnancy (suspected or diagnosed) or lactation;
* Use of disallowed concomitant therapy;
* History or suspicion of drug or alcohol abuse;
* Participation in an investigational drug trial within the 30 days prior to selection;
* Exhibits a disorder that is a contraindication to steroid hormonal therapy, including, for example, the following conditions:
* History of, or actual, thrombophlebitis or thromboembolic disorders;
* History of, or actual, cerebrovascular disorders;
* History of, or actual, myocardial infarction or coronary artery disease;
* Acute liver disease;
* History of, or actual, benign or malignant liver tumors;
* Known, or suspected, carcinoma of the breast;
* Known, or suspected, estrogen-dependent neoplasia;
* Undiagnosed abnormal vaginal bleeding;
* Any ocular lesion arising from opthalmic vascular disease, such as partial or complete loss of vision or defect in visual fields.
* Latex allergy.

Ages: 18 Years to 35 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 45
Dates: Start 2002-02; Study Completion 2002-12

PRIMARY OUTCOMES:
follicle growth
ovulation/anovulation
estradiol concentration
LH concentration

SECONDARY OUTCOMES:
endometrial development

CONTACTS AND LOCATIONS:
Overall Officials: Roger A Pierson, MS PhD, Principal Investigator — University of Saskatchewan
Locations (1):
- Ob-Gyn Royal University Hospital, Saskatoon, Saskatchewan, Canada

REFERENCES:
- [Background] Baerwald AR, Adams GP, Pierson RA. A new model for ovarian follicular development during the human menstrual cycle. Fertil Steril. 2003 Jul;80(1):116-22. doi: 10.1016/s0015-0282(03)00544-2. PMID 12849812
- [Background] Baerwald AR, Adams GP, Pierson RA. Characterization of ovarian follicular wave dynamics in women. Biol Reprod. 2003 Sep;69(3):1023-31. doi: 10.1095/biolreprod.103.017772. Epub 2003 May 14. PMID 12748128
- [Background] Pierson RA, Archer DF, Moreau M, Shangold GA, Fisher AC, Creasy GW. Ortho Evra/Evra versus oral contraceptives: follicular development and ovulation in normal cycles and after an intentional dosing error. Fertil Steril. 2003 Jul;80(1):34-42. doi: 10.1016/s0015-0282(03)00556-9. PMID 12849799